CLINICAL TRIAL: NCT05449522
Title: Effects of High Doses of Liquid Vitamin D Supplementation on Clinical Outcomes in Critically Traumatic Patients.
Brief Title: Vitamin D for Critically Traumatic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201705002MIPC
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Vitamin D Deficiency; Major Trauma
Keywords: Vitamin D; Major Trauma
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Experimental group will receive 576,000 IU on the 3rd post-trauma day and 432,000 IU on the 10th post-trauma day (1,008,000 IU in total) theoretically to achieve sufficient level of vitamin D.
  Interventions: Dietary Supplement: Vitamin D
- Control group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — High dose of vitamin D with 576,000 IU on the 3rd post-trauma day and 432,000 IU on the 10th post-trauma day (1,008,000 IU in total) is given orally or enterally via a feeding tube
  Arms: Treatment group
Dietary Supplement: Placebo — Medium-chain triglyceride (MCT)
  Arms: Control group

SUMMARY:
Trauma has been an important global public health issue. Yet it is the sixth cause of death in Taiwan, trauma brings great negative impact to national productivity since it presents specifically as the leading cause of death for the population aged below 40 years. According to the national databank from Formosa Association for the Surgery of Trauma, mortality rate in critically traumatic patients with injury severity score (ISS) ≥ 25 is as high as 23%. Vitamin D, a pleiotropic hormone, regulates directly functions of most organs and immune system. It has been proven that vitamin D insufficiency or deficiency would deteriorate survival of critically ill patients, while supplementation of high-dose vitamin D ameliorates the clinical outcomes. This study investigates whether multiple high doses of vitamin D supplementation in one week can decrease the mortality and morbidity in critically traumatic patients. The serum levels of calcidiol and PTH will be measured on Day 0, Day 3, Day 10, Day 15, Day 30 and Day 60 before and after vitamin D supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Major trauma adult (> 20 years old) with Injury Severity Score equal or higher than 9, who is admitted to ICU

Exclusion Criteria:

Patients with the following conditions:

* Chronic liver disease
* Contraindication to enteral feeds
* Hypercalcemia
* Current use of vitamin D, estrogen, or medications for bone disease
* High risk of hypercalcemia, ex. metastatic cancer, primary hyperparathyroidism, sarcoidosis, multiple myeloma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | up to 3 months after discharge
  Mortality in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Yi Han, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan